CLINICAL TRIAL: NCT05550883
Title: Effectiveness of Aerobic Exercises for Women With Fibromyalgia: a Randomized Controlled Trial
Brief Title: Aerobic Exercise for Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEFIBRO2022
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (aerobic exercise group) (Experimental): aerobic exercise training for 45 minutes, three sessions per week for 6 weeks.
  Interventions: Other: Aerobic exercise; Drug: Fibromyalgia Agents
- Group B (Medications group) (Active Comparator): The patients in this group did not receive treatment program. just received their medical treatment tricyclic antidepressants (low evening doses), and mostly when needed, low doses of: analgesics, muscle relaxants, hypnotics, and tranquilizers over the period of 6 weeks.
  Interventions: Drug: Fibromyalgia Agents

INTERVENTIONS:
Other: Aerobic exercise — The patients in this group participated in aerobic exercise training for 45 minutes, three sessions per week for 6 weeks. They underwent the proper warm up to minimize the risk of musculoskeletal injury .The training session started by a proper warm up for 5 min in the form of mild stretching for the involved muscle group to prepare the exercised muscles and improve blood supply for skeletal muscle to prevent fatigue or injury. Patients in this study group performed aerobic exercise (in the form of treadmill training) All sessions were supervised to ensure correct technique and monitor the appropriate amount of exercise. The training session ended by a proper cooling down for 5 min to prevent fatigue or injury.
  Arms: Group A (aerobic exercise group)
Drug: Fibromyalgia Agents — tricyclic antidepressants (low evening doses), and mostly when needed, low doses of: analgesics, muscle relaxants, hypnotics, and tranquilizers.

SUMMARY:
This is randomized controlled trial that investigated the effect of aerobic exercises in women with fibromyalgia. The study was performed in Abu-kabir central hospital - Al Sharquia, Egypt. The sample was recruited from the rheumatology department in Abu-kabir central hospital- Al Sharquia. Sixty women were included in the study based on the inclusion criteria. The first group (study group) included 30 participants who received aerobic exercise in addition to the prescribed medications. The second group (control group) included 30 participants who received the prescribed medications only. The outcome measures included visual analogue scale, Fibromyalgia Impact Questionnaire and cholesterol level. Assessment of outcomes were performed at baseline and after the end of treatment program.

ELIGIBILITY:
Inclusion Criteria:

* (1)Their ages ranged from 30 to 40 years old (2)Their body mass index (BMI) was from 20:26 kg/m2 (3)All patients assured diagnosis fibromyalgia for more than three months (4)Participants were on a stable regimen of pharmacological and/or non pharmacological treatment for FM the previous three months leading up to study period and agree to maintain their present medication unchanged for the duration of their participation in the study

Exclusion Criteria:

Patients with pregnancy, another accompanying central sensitization syndrome Patients with psychiatric illness Patients whose pharmacological treatment for FMS changed within the last three months Patients who do not have a cognitive level to answer the questions in the scale

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in Visual analogue scale | baseline and 6 weeks
  Visual Analaog Scale is used to measure the severity of pain in patients. The patient is told that there is no "0" pain on the 10 cm ruler drawn on paper, "10" is the most experienced pain, and the patient is asked to mark on the ruler according to the severity of the pain he/she feels. The distance of the marked point from zero is recorded as the Visual Analogue Scale score in cm.

SECONDARY OUTCOMES:
Changes in cholesterol level level | baseline and 6 weeks
  Blood sample to measure cholesterol level for each participant in both groups before and after treatment.
Changes in Fibromyalgia Impact Questionnaire | baseline and 6 weeks
  This questionnaire was designed to assess the current health status of patients with fibromyalgia. The FIQ has 11 individual questions and measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week ranging from 0-100 with higher score indicating more severity.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Abdeen, Ph.D, Principal Investigator — Cairo University
Locations (1):
- Abu-kabir central hosptial, Al Mansurah, Al Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided